CLINICAL TRIAL: NCT05553028
Title: Prospective Monocentric Randomized Study Comparing Arthrodesis Technique of Thoracic and/or Lumbar Spine by Posterior Approach Performed by Robot-assisted Surgery (Robot Mazor X Stealth ™) Versus Conventional Surgery
Brief Title: Study Comparing Arthrodesis Technique of Thoracic and/or Lumbar Spine by Posterior Approach Performed by Robot-assisted Surgery (Robot Mazor X Stealth ™) Versus Conventional Surgery
Acronym: ROBARTHRODESE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A00874-39
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Osteosynthesis; Mazor Robot; Spinal Surgery; Arthrosis; Spine
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot assisted surgery (Experimental): Patient operated for thoracic and/or lumbar spine arthrodesis with robot assistance Mazor
  Interventions: Procedure: Computerised tomography
- Conventional surgery (Active Comparator): Patient operated for thoracic and/or lumbar spine arthrodesis with conventional surgery
  Interventions: Procedure: Computerised tomography

INTERVENTIONS:
Procedure: Computerised tomography — Screws placement will be evaluated for each patient by a CT scan on D1 post-intervention. The evaluation of the placement of the screws (reading of the CT images) will be carried out by 2 radiologists independent of the surgical team, blinded to the technique used for the placement of the screws (robot-assisted/conventional surgery). In case of disagreement between the 2 evaluators, a 3rd evaluator will be requested.

SUMMARY:
Osteosynthesis by pedicle screwing is the reference technique since the 1980s, due to the quality of the mechanical grip of the screw in the pedicle, despite difficulties of placing the implant in this narrow tunnel.

This precision was improved by fluoroscopy, then by navigation, which made it possible to reduce the extra-pedicular placement of the screws and consequently the complications.

Since the 2000s, robotic has been developed in all areas, including medicine and surgery, (Da Vinci robot in urology) and several robots are currently marketed for spinal surgery, Medtronic's Mazor X Stealth ™ robot being the most successful.

The aim of this study is to evaluate on a prospective randomized comparative study the quality of the placement of the screws as well as the occurrence of complications, the clinical results and the medico-economic interest that robotic surgery can bring.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, over 18 years old,
* Any patient operated for thoracic and/or lumbar spine arthrodesis (spondylolisthesis, asymmetric disc disease, spinal instability, spinal deformities, advanced disc disease),
* Patient having given his free, informed and written consent to participate in the study,
* Patient able to answer questionnaires, able to communicate in the language of the country of the study,
* Negative pregnancy test,
* Patient affiliated to a social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Minor,
* Psychological disorders,
* Addiction to analgesics,
* Chronic infection,
* History of instrumented lumbar surgery,
* BMI greater than or equal to 40kg/m²,
* Pregnant or breastfeeding woman,
* Patient participating in another clinical study,
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of freedom by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of screw placement by a CT scan | one day
  Screws placement will be evaluated for each patient by a CT scan on D1 post-intervention. The evaluation of the placement of the screws (reading of the CT images) will be carried out by 2 radiologists independent of the surgical team, blinded to the technique used for the placement of the screws (robot-assisted/conventional surgery). In case of disagreement between the 2 evaluators, a 3rd evaluator will be requested.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint Martin, Pessac, France

REFERENCES:
- [Derived] Aurouer N, Guerin P, Cogniet A, Gangnet N, Pedram M, Piechaud PT; ReSurg; Mangione P. Pedicle screw placement accuracy in robot-assisted versus image-guided freehand surgery of thoraco-lumbar spine (ROBARTHRODESE): study protocol for a single-centre randomized controlled trial. Trials. 2024 Feb 3;25(1):106. doi: 10.1186/s13063-024-07908-1. PMID 38310274